CLINICAL TRIAL: NCT02205164
Title: Phase II Randomized Study of Multiple Doses of Palonosetron Plus Aprepitant Versus Multiple Doses of Palonosetron Alone in Preventing CINV in Patients With Newly Diagnosed AML or High-risk MDS Receiving Multiple Days Chemotherapy
Brief Title: Palonosetron Plus Aprepitant Versus Palonosetron in Preventing Nausea and Vomiting in Leukemic Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associazione Salentina Angela Serra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AS/PALO/002; 2011-003823-36 (EudraCT Number)
Record Dates: First submitted 2014-07-17; First posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
Keywords: palonosetron; aprepitant; CINV; AML; multiple-days
MeSH Terms: conditions — Vomiting | interventions — Palonosetron; Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palonosetron + Aprepitant (Experimental): Oral aprepitant will be given on days 1-3 (day 1, 125 mg 1 h before chemohterapy; days 2-3, 80 mg) multiple intravenous bolus of palonosetron 0.25 mg, 30 minutes before chemotherapy, every other single days, for a minimum of 2 administration (day 1, 3), in case of a 3 days chemotherapy regimen, and a maximum of 5 doses (day 1,3,5,7, 9) in case of a 10 days chemotherapy.
  Interventions: Drug: Palonosetron + Aprepitant
- Palonosetron (Active Comparator): multiple intravenous bolus of palonosetron 0.25 mg, 30 minutes before chemotherapy, every other single days, for a minimum of 2 administration (day 1, 3), in case of a 3 days chemotherapy regimen, and a maximum of 5 doses (day 1,3,5,7, 9) in case of a 10 days chemotherapy.
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Palonosetron + Aprepitant — Aloxi 0.25mg Emend 125/80/80 mg
  Other Names: Aloxi + Emend
  Arms: Palonosetron + Aprepitant
Drug: Palonosetron — Aloxi 0.25mg
  Other Names: Aloxi
  Arms: Palonosetron

SUMMARY:
The aim of present study is to evaluate if the addition of Aprepitant to multiple doses of palonosetron IV enhances the efficacy of multiple doses of palonosetron IV alone, in preventing CINV in AML or High risk MDS patient, treated with multiple days chemotherapy.

DETAILED DESCRIPTION:
This is an open-label, randomized, comparative, multicenter phase II study in patients with AML scheduled to receive multiple days chemotherapy.

Patients will receive either PALO+APR or the PALO regimen in a 1:1 ratio according to a computer-generated, random allocation schedule. Below are described the details for both antiemetic regimens:

PALO+APR regimen: oral aprepitant will be given on days 1-3 (day 1, 125 mg, days 2-3, 80 mg 1 hour before chemotherapy ) and multiple intravenous bolus of Palonosetron without dexamethasone, prior to the administration of chemotherapy, starting the first day of treatment.

PALO regimen: multiple intravenous bolus of Palonosetron without dexamethasone, prior to the administration of chemotherapy, starting the first day of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Myeloid Leukaemia or High-risk MDS according to IPSS
* Patient eligible for AML-like induction therapy
* Candidate for multiple-days chemotherapy (minimum 3 days)
* Age more, equal18 years
* ECOG 0-2
* Not pregnant or nursing
* Must be able to complete the patient's diary
* Provide written informed consent

Exclusion Criteria:

* AML or HR-MDS therapy-related
* Active infection requiring intravenous antibiotics
* Prior malignancies at other sites except surgically treated non-melanoma skin cancer, prostate cancer, superficial cervical cancer, or other cancer from which the patient had been disease-free for more/equal 5 years
* Unacceptable hepatic function (more of 2 times the upper limit of normal for liver transaminases) and renal function (creatinine more of 1.5 times the upper limit of normal) unless disease-related
* Myocardial infarction within the past 6 months
* Psychiatric or CNS disorders interfering with ability to comply with study protocol
* Known hypersensitivity to 5-HT3 antagonists and their components CSF involvement
* Pre-existing nausea or vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Complete Response | 5 days after chemotherapy
  The primary endpoint is the overall rate of patients achieving a complete response (defined as no emetic episode and no use of rescue medication) during the overall phase.

SECONDARY OUTCOMES:
Complete Control | 5 days after chemotherapy
  No emetic episode, no need for rescue medication, with a maximum grade of mild nausea
Emesis-free | 5 days after chemotherapy
  Percentage of patients without emetic episodes
Presence of nausea | 5 days after chemotherapy
  Presence of nausea graded according to Likert scale (none, mild, moderate and severe)
Treatment failure | 5 days after chemotherapy
  Time (days) to treatment failure (first emetic episode or first need of rescue medication, whichever occurs first)
Patient global satisfaction | 5 days after chemotherapy
  Patient global satisfaction with antiemetic therapy, as measured by a visual analogue scale (VAS)
Safety and tolerability | 5 days after chemotherapy
  Number of patients experienced at least one adverse events related to study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Di Renzo, MD, Principal Investigator — Ospedale Vito Fazzi
Locations (11):
- Italy (11):
  - Università-Azienda Policlinico di Bari, Bari, BA
  - Ospedale Perrino, Brindisi, BR
  - Ospedale Pugliese-Ciacco, Catanzaro, CZ
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - Ospedale Vito Fazzi, Lecce, LE
  - Ospedale "Cardinale Panico", Tricase, LE
  - A.O. Riuniti Papardo - Piemonte, Messina, ME
  - Casa di Cura "La Maddalena", Palermo, PA
  - Ospedale Ascoli Civico Palermo, Palermo, PA
  - Ospedale Moscati, Taranto, TA
  - ARON " Cardarelli", Napoli

REFERENCES:
- [Derived] Di Renzo N, Melillo L, Porretto F, Dargenio M, Pavone V, Pastore D, Mazza P, Mannina D, Merenda A, Cascavilla N, Greco G, Matera R, Bonizzoni E, Celio L, Musso M. Every-other-day palonosetron plus aprepitant for prevention of emesis following induction chemotherapy for acute myeloid leukemia: A randomized, controlled study from the "Rete Ematologica Pugliese". Cancer Med. 2020 Jan;9(1):170-178. doi: 10.1002/cam4.2628. Epub 2019 Nov 14. PMID 31725196